CLINICAL TRIAL: NCT05771389
Title: Correlation of RAFTLIN-1 Levels and Clinical Parameters in Axial Spondyloarthritis and Psoriatic Arthritis
Brief Title: RAFTLIN-1 Levels in Axial Spondyloarthritis and Psoriatic Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 17.11.2021-E.40188
Record Dates: First submitted 2023-03-05; First posted 2023-03-16 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Axial Spondyloarthritis; Psoriatic Arthritis
Keywords: Axial Spondyloarthritis; Psoriatic Arthritis; Raftlin-1
MeSH Terms: conditions — Axial Spondyloarthritis; Arthritis, Psoriatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Psoriatic arthritis (Active Comparator): Patients meeting the CASPAR (ClASsification criteria for Psoriatic ARthritis) criteria
  Interventions: Diagnostic Test: serum raftlin-1 protein levels
- Axial spondyloarthritis (Active Comparator): Patients meeting the ASAS classification criteria for axial spondyloarthritis
  Interventions: Diagnostic Test: serum raftlin-1 protein levels
- Healthy controls (Placebo Comparator): Healthy people who do not have inflammatory conditions.
  Interventions: Diagnostic Test: serum raftlin-1 protein levels

INTERVENTIONS:
Diagnostic Test: serum raftlin-1 protein levels — Lipid raft linker 1 (Raftlin-1) is a protein which enables double-stranded RNA binding activity. It is involved in T cell receptor signaling pathway; membrane raft assembly; and positive regulation of growth rate. It acts upstream of or within dsRNA transport; response to exogenous dsRNA; and toll-like receptor signaling pathway. Located in endosome; membrane raft; and plasma membrane.

SUMMARY:
Unlike other rheumatic diseases, acute phase reactants such as C-reactive protein and erythrocyte sedimentation rate are not diagnostic for patients with Spondyloarthropathies (SpA). Also, it is not possible to monitor disease activity with these tests. On the other hand, HLA-B27 positivity varies between races, and 8% of the normal population is HLA-B27 positive. In this manner, new biomarkers for endorsing the diagnosis and monitoring the disease activity are necessary.

Acute phase reactants are not sensitive for diagnosing and assessing disease activity. This may lead to a diagnostic delay of up to 9 years. The investigators hypothesize that Raftlin-1, thought to have a regulatory role in TH17 function and IL-17-mediated immunity, may be a novel biomarker for showing inflammation-related clinical features.

DETAILED DESCRIPTION:
Unlike other rheumatic diseases, acute phase reactants such as C-reactive protein and erythrocyte sedimentation rate are not diagnostic for patients with Spondyloarthropathies (SpA). Also, it is not possible to monitor disease activity with these tests. On the other hand, HLA-B27 positivity varies between races, and 8% of the normal population is HLA-B27 positive. In this manner, new biomarkers for endorsing the diagnosis and monitoring the disease activity are necessary.

In recent years Raftlin, a significant lipid raft protein responsible for transmembrane signal transmission, was found. It has been discovered that the Raftlin protein has two subtypes (Raftlin-1 and Raftlin-2), and in transgenic mice without RAFTLIN genes, T-cell-dependent immunity has been altered.

Cytokine production, especially IL-17, is diminished in T cells with the lack of Raftlin protein, while it is increased in T cells, including transgenic Raftlin. This condition is associated with TCR-related signaling pathways. Particularly, Lck protein occurrence in lipid raft is increased with Raftlin overexpression, while it is diminished with absence. Regarding this, Raftlin is thought to modulate TCR signaling, thus altering the T-cell mediated immunity.

Acute phase reactants are not sensitive for diagnosing and assessing disease activity. This may lead to a diagnostic delay of up to 9 years. The investigators hypothesize that Raftlin-1, thought to have a regulatory role in TH17 function and IL-17-mediated immunity, may be a novel biomarker for showing inflammation-related clinical features.

ELIGIBILITY:
Inclusion Criteria:

* Being aged 18 to 65
* Meeting ASAS axial spondyloarthritis classification criteria
* Meeting The CASPAR (ClASsification criteria for Psoriatic ARthritis) criteria

Exclusion Criteria:

* Having a burn or a wound
* Active infection
* systemic inflammatory disease (Type 1 DM, autoimmune thyroiditis, other inflammatory rheumatic conditions etc.)
* Pregnancy
* Malignancy
* severe cognitive function disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2023-07-09 (Actual); Study Completion 2023-07-09 (Actual)

PRIMARY OUTCOMES:
Bath Ankylosing Spondylitis Disease Activity Index(BASDAI) | 1 day
  This questionnaire evaluates the disease activity level in patients with AS. The BASDAI consists of a 0 - 10 scale measuring discomfort, pain, and fatigue (0 being no problem and 10 being the worst problem) in response to six questions asked of the patient pertaining to the five major symptoms of AS. The final score varies between 0 and 10.
Bath Ankylosing Spondylitis Disease Activity Index(BASFI) | 1 day
  This questionnaire evaluates the functionality in patients with AS. The ten questions that comprise the BASFI were chosen with input from patients with AS. The first 8 questions evaluate activities related to functional anatomical limitations due to the course of this inflammatory disease. The final 2 questions evaluate the patients' ability to cope with everyday life. A visual analogue scale (with 0 being "easy" and 10 "impossible) is used to answer the questions on the test. The final score varies between 0 and 10.
The Ankylosing Spondylitis Disease Activity Score (ASDAS) | 1 day
  AS Disease Activity Score has been developed by taking into account total back pain (Bath Ankylosing Spondylitis Disease Activity Index [BASDAI] question 2), patient global evaluation, peripheral joint pain or swelling (BASDAI question 3), duration of morning stiffness (BASDAI question 6), and C-reactive protein (CRP) (or erythrocyte sedimentation rate [ESR] if CRP is not available). The cutoffs between the disease activity states are inactive disease ≤1.3, moderate 1.3-2.0, high 2.1-3.5, and very high ≥3.5. The ASDAS cutoff for clinically important improvement between examinations is ≥1.1, and the cutoff for a major improvement is ≥2.0.
Bath Ankylosing Spondylitis Metrology Index(BASMI) | 1 day
  Bath Ankylosing Spondylitis Metrology Index, a combined index to assess the spinal mobility. It evaluates the patients regarding cervical rotation, tragus-to-wall distance, lumbar flexion, lumbar lateral flexion and intermalleolar distance. The total score varies between 5 to 15 in patients with ankylosing spondylitis
Disease Activity Index for Psoriatic Arthritis (DAPSA) | 1 day
  DAPSA includes a 68/66 joint count summed with a patient global, patient pain score, and C- reactive protein level. The DAPSA provides a continuous score of arthritis activity and has validated cut points for remission (< 4) and low disease activity (< 14).
Spondyloarthritis Research Consortium of Canada Enthesitis Index(SPARCC Enthesitis Index) | 1 day
  The Spondyloarthritis Research Consortium of Canada (SPARCC) index, developed in Canada by Walter Maksymowych and others, was developed in patients with spondyloarthritis and includes assessment of 18 sites for tenderness. The total score is 16, because the distal patella and tibial tuberosity, in close proximity, are considered as one site. The core is between 0 and 16.
Health Assessment Questionnaire (HAQ) | 1 day
  The Health assessment questionnaire (HAQ) is a questionnaire for the assessment of disability in an individual. The patients report the amount of difficulty they have in performing eight daily living activities. Each question asks on a scale ranging from 0 to 3 if the categories can be performed without any difficulty (scale 0) up to cannot be done at all (scale 3). The final score varies between 0 and 3.
numeric rating scale (rest, movement) | 1 day
  Self reported pain scored between 0 (minimum)-10 (maximum). Higher scores represent a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ozan Volkan Yurdakul, Assoc. Prof., Principal Investigator — Bezmialem University; Mert Kara, MD, Principal Investigator — Bezmialem University; Ömer Faruk Özer, Assoc. Prof., Principal Investigator — Bezmialem University
Locations (1):
- Bezmialem University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rudwaleit M, Haibel H, Baraliakos X, Listing J, Marker-Hermann E, Zeidler H, Braun J, Sieper J. The early disease stage in axial spondylarthritis: results from the German Spondyloarthritis Inception Cohort. Arthritis Rheum. 2009 Mar;60(3):717-27. doi: 10.1002/art.24483. PMID 19248087
- [Background] Saeki K, Miura Y, Aki D, Kurosaki T, Yoshimura A. The B cell-specific major raft protein, Raftlin, is necessary for the integrity of lipid raft and BCR signal transduction. EMBO J. 2003 Jun 16;22(12):3015-26. doi: 10.1093/emboj/cdg293. PMID 12805216
- [Background] Saeki K, Fukuyama S, Ayada T, Nakaya M, Aki D, Takaesu G, Hanada T, Matsumura Y, Kobayashi T, Nakagawa R, Yoshimura A. A major lipid raft protein raftlin modulates T cell receptor signaling and enhances th17-mediated autoimmune responses. J Immunol. 2009 May 15;182(10):5929-37. doi: 10.4049/jimmunol.0802672. PMID 19414744
- [Derived] Yurdakul OV, Kara M, Ince B, Yildiz C, Yildiz T, Kilicoglu MS, Aydin T, Ozer OF. Raftlin - a potential biomarker for axial spondyloarthritis and psoriatic arthritis: An observational study. Medicine (Baltimore). 2024 Jun 28;103(26):e38770. doi: 10.1097/MD.0000000000038770. PMID 38941376